CLINICAL TRIAL: NCT01588015
Title: A Phase I Trial to Evaluate Safety and Immunogenicity of a Cytomegalovirus Peptide Vaccine Co-Injected With PF-03512676 Adjuvant in Recipients of Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: Vaccine Therapy in Preventing Cytomegalovirus Infection in Patients With Hematological Malignancies Undergoing Donor Stem Cell Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12022; NCI-2012-00589 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Promyelocytic Leukemia (M3); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Adult Nodular Lymphocyte Predominant Hodgkin Lymphoma; Anaplastic Large Cell Lymphoma; B-cell Adult Acute Lymphoblastic Leukemia; Chronic Eosinophilic Leukemia; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Contiguous Stage II Adult Burkitt Lymphoma; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Lymphoblastic Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cytomegalovirus Infection; de Novo Myelodysplastic Syndromes; Essential Thrombocythemia; Extramedullary Plasmacytoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Isolated Plasmacytoma of Bone; Monoclonal Gammopathy of Undetermined Significance; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Peripheral T-cell Lymphoma; Polycythemia Vera; Post-transplant Lymphoproliferative Disorder; Previously Treated Myelodysplastic Syndromes; Primary Central Nervous System Hodgkin Lymphoma; Primary Central Nervous System Non-Hodgkin Lymphoma; Primary Myelofibrosis; Progressive Hairy Cell Leukemia, Initial Treatment; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Stage I Adult Burkitt Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Lymphoblastic Lymphoma; Stage I Adult T-cell Leukemia/Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Cutaneous T-cell Non-Hodgkin Lymphoma; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Multiple Myeloma; Stage I Small Lymphocytic Lymphoma; Stage IA Mycosis Fungoides/Sezary Syndrome; Stage IB Mycosis Fungoides/Sezary Syndrome; Stage II Adult Hodgkin Lymphoma; Stage II Adult T-cell Leukemia/Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Cutaneous T-cell Non-Hodgkin Lymphoma; Stage II Multiple Myeloma; Stage IIA Mycosis Fungoides/Sezary Syndrome; Stage IIB Mycosis Fungoides/Sezary Syndrome; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Adult T-cell Leukemia/Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Cutaneous T-cell Non-Hodgkin Lymphoma; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Multiple Myeloma; Stage III Small Lymphocytic Lymphoma; Stage IIIA Mycosis Fungoides/Sezary Syndrome; Stage IIIB Mycosis Fungoides/Sezary Syndrome; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Adult T-cell Leukemia/Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Cutaneous T-cell Non-Hodgkin Lymphoma; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Small Lymphocytic Lymphoma; Stage IVA Mycosis Fungoides/Sezary Syndrome; Stage IVB Mycosis Fungoides/Sezary Syndrome; T-cell Adult Acute Lymphoblastic Leukemia; T-cell Large Granular Lymphocyte Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Hairy Cell Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Promyelocytic, Acute; Lymphoma, Extranodal NK-T-Cell; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Cytomegalovirus Infections; Thrombocythemia, Essential; Monoclonal Gammopathy of Undetermined Significance; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Polycythemia Vera; Primary Myelofibrosis; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (vaccine therapy) (Experimental): Patients receive Tet-CMV + PF03512675 SC on days 28 and 56 post-HCT.
  Interventions: Biological: tetanus-CMV fusion peptide vaccine; Other: laboratory biomarker analysis
- Arm II (control) (Active Comparator): Patients undergo immune monitoring only.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: tetanus-CMV fusion peptide vaccine — Given SC
  Arms: Arm I (vaccine therapy)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase I trial studies the side effects of vaccine therapy in preventing cytomegalovirus (CMV) infection in patients with hematological malignancies undergoing donor stem cell transplant. Vaccines made from a tetanus-CMV peptide or antigen may help the body build an effective immune response and prevent or delay the recurrence of CMV infection in patients undergoing donor stem cell transplant for hematological malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To discover whether two administrations of 2.5 mg tetanus (Tet)-CMV peptide co-injected with 1 mg of PF-03512676 (tetanus-CMV fusion peptide vaccine), by subcutaneous (SC) route on days 28 and 56 post-hematopoietic cell transplantation (HCT) are safe and well tolerated in human leukocyte antigen (HLA) A*0201 CMV-positive recipients of allogeneic HCT.

SECONDARY OBJECTIVES:

I. To measure levels of CMV-specific T cells in vaccinated compared to unvaccinated HCT recipients (control arm).

II. To assess whether vaccination of HCT recipients with Tet-CMV co-injected with PF03512676 reduces expression of programmed death 1 (PD-1) on CMV-specific T cells.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive Tet-CMV + PF03512675 SC on days 28 and 56 post-HCT.

ARM II: Patients undergo immune monitoring only.

After completion of study treatment, patients are followed up at days 70, 84, 100, 130, 160, and 180.

ELIGIBILITY:
Inclusion Criteria:

* HLA A*0201 subtype
* CMV seropositive
* Able and willing to sign the informed consent form (ICF)
* Willingness to be followed for the planned duration of the trial (6 months post-HCT)
* Seronegative for human immunodeficiency virus (HIV), hepatitis C virus (HCV) and active hepatitis B virus (HBV) (surface antigen negative)
* Planned related or unrelated HCT, with 8/8 or 7/8 (A, B, C, DRB1) high resolution HLA donor allele matching
* HCT for the treatment of hematologic cancers including, but not limited to:

  * Acute lymphoblastic leukemia in first or second remission (for acute lymphoblastic leukemia/lymphoblastic lymphoma, the disease status needs to be in hematologic remission by bone marrow/peripheral blood; persistent lymphadenopathy on computed tomography [CT] or CT/positron emission tomography [PET] scan without progression is allowed)
  * Chronic myelogenous leukemia in first chronic or accelerated phase, or in second chronic phase
  * Hodgkin and non-Hodgkin lymphoma
  * Myelodysplastic syndrome
* Planned HCT with minimal to no-T cell depletion of graft
* Use of contraception up to 90 days post-HCT
* Negative pregnancy test for female recipient
* DISEASE STATUS: Recipients to be enrolled are patients eligible for allogeneic HCT, who were diagnosed with hematologic cancers including:
* Acute lymphoblastic leukemia (ALL); B-precursor ALL; T cell ALL
* Acute myeloid leukemia (AML), acute promyelocytic leukemia; treatment related AML
* Chronic lymphoid leukemia; adult T cell leukemia/lymphoma, chronic lymphocytic leukemia not otherwise specified (NOS), hairy cell leukemia; prolymphocytic leukemia (B or T); T cell large granular (gran.) lymphocytic (lymph.) leukemia (leuk)
* Chronic myeloproliferative disease (CML); chronic eosinophilic leukemia (CEL)/hypereosinophilic syndrome; chronic idiopathic myelofibrosis; CML - Philadelphia chromosome; essential thrombocythemia; polycythemia vera
* Leukemia, not otherwise specified (NOS)
* Myelodysplastic syndrome, NOS; chronic myelomonocytic leukemia
* Hodgkin lymphoma, NOS; Hodgkin lymphoma nodular lymphocyte predominant (LP), NOS; Hodgkin lymphoma - like post-transplant lymphoproliferative disorder (PTLD)
* Lymphoma, NOS
* Non-Hodgkin lymphoma (NHL); anaplastic large-cell lymphoma (ALCL), cutaneous, ALCL, systemic; Burkitt lymphoma/leukemia; cutaneous T-cell lymphoma (CTCL)/mycosis fungoides; CTCL/Sezary syndrome; diffuse large B-cell lymphoma; mucosa associated lymphoid tissue (MALT)-lymphoma; extranodal natural killer (NK)/T cell lymphoma, extranodal NK/T lymphoma nasal; follicular lymphoma; lymphoplasmacytic lymphoma mantle cell lymphoma; mediastinal large B-cell lymphoma; nodal marginal zone B-cell lymphoma (lymph.); NHL aggressive, NOS; NHL indolent, NOS; NHL, NOS; peripheral T cell lymphoma, NOS; PTLD (monoclonal); PTLD (polyclonal); precursor (precur.) B-lymphoblastic lymphoma; precur T-lymphoblastic lymphoma; primary central nervous system (CNS) lymphoma; primary effusion lymphoma; small lymphocytic lymphoma, NOS
* Myeloma, NOS; monoclonal gammopathy of undetermined significance (MGUS); solitary plasmacytoma
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately
* All medications, supportive care, blood products or radiation therapy taken or administered during the trial will be documented in the subject's clinical/hospital and case report form (CRF), using City of Hope (COH) guidelines; the subject's clinical information will be recorded on the appropriate CRF
* Concurrent enrollment in other clinical trials using an investigational product is prohibited
* The use of alemtuzumab for immunosuppression is not permitted in this study
* Prophylactic therapy with CMV immunoglobulin or prophylactic antiviral CMV treatment is not allowed
* Medications that might interfere with the evaluation of the investigational product should not be administered, from 30 days prior to participation on the trial and up to 14 days after the second vaccination (day 70 post-HCT); medications in this category include, but are not limited to:

  * Live attenuated vaccines
  * Medically indicated subunit (Engerix-B for HBV; Gardasil for HPV) or killed vaccines (e.g. influenza, pneumococcal, or allergy treatment with antigen injections)
* Antiviral treatment for herpes simplex virus (HSV), human herpes virus 6 (HHV6), Epstein-Barr virus (EBV) and adenovirus including the use of GVC/VAL, FOS, Cidofovir, CMX-001 may also suppress reactivation of CMV, thus it will not be allowed in this study; patients requiring such treatment before randomization (day 28) will be removed from the study and replaced; reasons for removal will be reported in the patient's CRF
* All enrolled recipients who will require anti-CMV therapy before day 28 will be replaced, treated and monitored as required by COH standard of care; GVC/VAL, FOS, Cidofovir, CMX-001 may be used according to COH standard of care (SOC) for preemptive management of CMV viremia; should antiviral treatment be required after day 28, the planned 2nd vaccine injection at day 56 will not be administered (vaccine arm only)
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* A poor-risk patient, as defined by any of the following:

  * Chronic myelogenous leukemia in blast crisis
  * Acute myeloid leukemia beyond second remission
  * Multiple myeloma
  * Aplastic anemia
* Planned immunosuppression with alemtuzumab or any equivalent in vivo T-cell depleting agent
* In vitro T cell depleted graft
* Planned prophylactic therapy with CMV immunoglobulin
* Planned CMV prophylactic therapy
* Experimental anti-CMV chemotherapy in the last 6 months
* Diagnosed with autoimmune disease
* Receipt of the following substances:

  * Any prior investigational CMV vaccine
  * Live attenuated vaccines, medically indicated subunit or killed vaccines from 30 days prior to participation in the trial and up to 14 days after the second vaccination (day 70 post-HCT)
  * Investigational research products or allergy treatment with antigens injections from 30 days prior to participation in the trial and up to 14 days after the second vaccination (day 70 post-HCT)
* Pregnant and/or breast feeding if a female recipient
* Refusing to use contraception up to 90 days post-HCT
* POST-HCT STUDY-SPECIFIC EXCLUSIONS:
* On days 28 and 56 post-HCT (immunization day for the vaccine arm) all study recipients (vaccine and observation arms) will be reviewed for eligibility and ruled ineligible to initiate or continue in the study and receive vaccination (for the vaccine arm) if:

  * Diagnosed with > grade 2 graft-versus-host disease (GVHD) before day 28 post-HCT, and diagnosed with > grade 2 GVHD between day 28 post-HCT and administration of the 2nd vaccine at day 56
  * Received steroid therapy with prednisone > 1 mg/kg/day, less than 7 days prior to injection
  * Had relapse
  * Experience graft failure (absolute neutrophil count < 500/mm^3)
  * Received antiviral treatment with GVC/VAL, FOS, Cidofovir, CMX-001 at any point during the 28 day period
  * There are ongoing non-hematological post-HCT toxicities >= grade 3 non-hematological (hem) adverse events (AE's), with exception of grade 3 glucose intolerance and grade 3 non-hem labs; cholesterol, triglyceride, and hyperglycemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10-29 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Safety based on assessment of GVHD, graded according to the Keystone Consensus system and adverse events (AEs) based on National Cancer Institute (NCI) CTCAE version 4.03 | Up to day 180
  GVHD, local and systemic reactogenicity, and toxicity related to the vaccine formulation will be evaluated by the study principal investigator (PI), conferring with the treating physician. AEs will be summarized for each treatment group by type (MedDRA codes within organ systems), grade, and attribution.

SECONDARY OUTCOMES:
Immunogenicity evaluated by monitoring CMV-specific CD8+ T cells by multi color flow cytometric analyses | Up to day 180
  Compare levels of CD8+ T cells binding to CMV-specific tetramers in vaccinated and unvaccinated HCT recipients by Wilcoxon rank-sum test, using integrated CMV-specific CD8+ T cells levels over the first 100 days as a numerical outcome. PD-1 expression and levels of apoptosis markers and proliferation of CMV-specific T cells immune-parameters will be compared in both arms using the Kruskall-Wallis rank-sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Ryotaro Nakamura, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] La Rosa C, Longmate J, Lingaraju CR, Zhou Q, Kaltcheva T, Hardwick N, Aldoss I, Nakamura R, Diamond DJ. Rapid Acquisition of Cytomegalovirus-Specific T Cells with a Differentiated Phenotype, in Nonviremic Hematopoietic Stem Transplant Recipients Vaccinated with CMVPepVax. Biol Blood Marrow Transplant. 2019 Apr;25(4):771-784. doi: 10.1016/j.bbmt.2018.12.070. Epub 2018 Dec 16. PMID 30562587
- [Derived] Nakamura R, La Rosa C, Longmate J, Drake J, Slape C, Zhou Q, Lampa MG, O'Donnell M, Cai JL, Farol L, Salhotra A, Snyder DS, Aldoss I, Forman SJ, Miller JS, Zaia JA, Diamond DJ. Viraemia, immunogenicity, and survival outcomes of cytomegalovirus chimeric epitope vaccine supplemented with PF03512676 (CMVPepVax) in allogeneic haemopoietic stem-cell transplantation: randomised phase 1b trial. Lancet Haematol. 2016 Feb;3(2):e87-98. doi: 10.1016/S2352-3026(15)00246-X. Epub 2015 Dec 24. PMID 26853648